CLINICAL TRIAL: NCT02316743
Title: Beneficial Effects of Levothyroxine Supplementation in Patients With Systolic Heart Failure and Subclinical Hypothyroidism
Brief Title: Effects of Levothyroxine Supplementation in Patients With Systolic Heart Failure and Subclinical Hypothyroidism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Paul Farand, Investigator, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thyroid-001
Record Dates: First submitted 2013-05-10; First posted 2014-12-15 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Systolic Heart Failure; Sub-clinical Hypothyroidism
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levothyroxine (Experimental): Levothyroxine supplementation
  Interventions: Drug: Levothyroxine supplementation

INTERVENTIONS:
Drug: Levothyroxine supplementation — T4 supplementation for heart failure patients with subclinical hypothyroidism.
  Other Names: T4 supplementation

SUMMARY:
The purpose of this study is to determine whether levothyroxine supplementation is beneficial in patients with systolic heart failure and subclinical hypothyroidism on the functional class evaluated with a 6 minute walk test.

DETAILED DESCRIPTION:
Forty patients with systolic heart failure and subclinical hypothyroidism will be include in a open label trial. They will receive levothyroxine supplementation to determine if their functional class will be affect.

ELIGIBILITY:
Inclusion Criteria:

* Biochemical diagnosis of subclinical hypothyroidism (TSH between 3.5 and 10 with a normal T4)
* Systolic heart failure with New-York Heart Association (NYHA) class II or III
* Left ventricular ejection fraction under 40%
* Stable heart failure for the past 3 months (no IV furosemide or hospital admission)
* Beta-blockers and ACE inhibitors titrated to the maximum tolerated dose

Exclusion Criteria:

* Isolated diastolic heart failure
* Awaiting cardiac resynchronisation therapy
* Impossibility to perform the 6 minutes walk test
* Active cancer / Life expectancy under 18 months
* Treatment with amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Performance at the 6 minutes walk test | 6 months

SECONDARY OUTCOMES:
Difference of the brain natriuretic peptide measurement | 6 months
Difference of activin a measurement | 6 months
Difference of myostatin measurement | 6 months
Increase in heart rate measurement | 6 months
  Absence / Presence of tachycardia (heart rate > 100 beat per minute) at baseline and 6 months
Difference of systolic and diastolic function on transthoracic echocardiogram | 6 months
Arhythmic (ventricular arrhythmias and supraventricular arrythmias) and ischemic events (myocardial infarction, unstable angina and hospitalization for revascularization) | 6 months
Normalisation of thyroid workup | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel Nguyen, MD, Study Director — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada